CLINICAL TRIAL: NCT01354535
Title: Isolated Locked Compression Plating Versus Cable Plating and Strut Allografts With Cerclage Wiring for Vancouver B1 Periprosthetic Femoral Fractures: A Randomized Controlled Trial
Brief Title: Types of Fixation of Vancouver B1 Periprosthetic Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13052011
Record Dates: First submitted 2011-05-13; First posted 2011-05-17 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Femur Fractures
Keywords: periprosthetic; femur fractures; Vancouver B1
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cable plating with strut (Active Comparator): The plate will be placed laterally with the allograft strut placed on the anterior cortex. Screw fixation will be used distal to the stem and cables and screws will be used proximal to the stem tip. Cerclage cables or wires will be used to secure the strut.
  Interventions: Procedure: Cable Plating and Strut Allograft with Cerclage Wiring
- isolated plating (Active Comparator): A lateral thigh incision will be used to expose the fracture site. Surgeons will attempt to minimize devascularization of the bone by meticulous dissection and indirect reduction techniques. An appropriate sized plate will be applied to the lateral aspect of the femur. Fracture reduction will be achieved with the use of intra-operative fluoroscopy and the plate will be secured with locking screws.
  Interventions: Procedure: Isolated Locked Compression Plate

INTERVENTIONS:
Procedure: Isolated Locked Compression Plate — A lateral thigh incision will be used to expose the fracture site. Surgeons will attempt to minimize devascularization of the bone by meticulous dissection and indirect reduction techniques. An appropriate sized plate will be applied to the lateral aspect of the femur. Fracture reduction will be achieved with the use of intra-operative fluoroscopy and the plate will be secured with locking screws.
  Arms: isolated plating
Procedure: Cable Plating and Strut Allograft with Cerclage Wiring — The plate will be placed laterally with the allograft strut placed on the anterior cortex. Screw fixation will be used distal to the stem and cables and screws will be used proximal to the stem tip. Cerclage cables or wires will be used to secure the strut.
  Arms: Cable plating with strut

SUMMARY:
The purpose of this study is to compare two different but standard treatments for the fixation of Vancouver B1 periprosthetic. The investigators aim to compare open reduction internal fixation using a locked plating system versus plating and strut allograft with cerclage wiring to determine which treatment results in a faster return to function as measured by the TUG test at 6 weeks post-op.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18, no upper limit
* Vancouver type B1 periprosthetic fracture
* Fracture is amenable to either treatment group
* Prosthesis is well fixed
* Provision of informed consent

Exclusion Criteria:

* Presence of an active infection around the fracture (soft tissue or bone)
* Loose prosthesis
* Trauma patients with an ISS > 16 or associated major injuries of the lower extremities
* Known substance abuse
* Likely problems, in the judgment of the investigators, with maintaining follow-up (i.e., patients with no fixed address, report a plan to move out of town, or intellectually challenged patients without adequate family support)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2013-02; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
TUG test score at 6 weeks post-op | 6 weeks
  We will administer the TUG test to each patient at 6 weeks to determine if there is a difference in functional status between both groups.

SECONDARY OUTCOMES:
Re-operation rates | 1 year
  We will measure rates of re-operationin each of the treatment groups on study specific case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Schemitsch, MD, FRCS(C), Principal Investigator — Unity Health Toronto; Aaron Nauth, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. michael's Hospital, Toronto, Ontario, Canada